CLINICAL TRIAL: NCT05335252
Title: Dronabinol for the Treatment of Postoperative Pain After Arthroscopic Surgery: a Pilot Randomized Trial
Brief Title: Dronabinol After Arthroscopic Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Vehniah Tjong, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00213383
Record Dates: First submitted 2022-04-13; First posted 2022-04-19 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis; Knee Injuries; Meniscus Tear; Synovitis of Knee; Knee Ligament Injury; Chondral Injury of Left Knee; Chondral Injury of Right Knee; Loose Body Knee
Keywords: Knee Arthroscopy
MeSH Terms: conditions — Osteoarthritis, Knee; Knee Injuries | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dronabinol (Experimental): Patients will received dronabinol (5mg) twice a day for 7 days in addition to standard pain medication protocol after arthroscopic knee surgery
  Interventions: Drug: Dronabinol
- Placebo (Placebo Comparator): Patients will received placebo twice a day for 7 days in addition to standard pain medication protocol after arthroscopic knee surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — 5mg 2x daily for 7 days
  Other Names: Marinol
  Arms: Dronabinol
Drug: Placebo — 1 caplet 2x daily for 7 days
  Arms: Placebo

SUMMARY:
The purpose of the proposed study is to evaluate the efficacy of dronabinol for postoperative pain after arthroscopic surgery of the knee. The investigators hypothesize that dronabinol will relieve pain, reduce opioid consumption and will result in few negative side effects. If this pilot study shows promising results the investigators will expand the trial to include additional arthroscopic surgeries (hip, shoulder) and other types of orthopaedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patient who will undergo arthroscopic surgery of the knee including, but not limited to,

  * Meniscectomy
  * Synovectomy
  * Chondroplasty
  * Loose body removal

Exclusion Criteria:

* Patients under age 18 years
* Patients who cannot provide consent
* Patients who are pregnant, breast feeding, or are trying to become pregnant during the study period
* Patients with an allergy to any of the study drugs
* Patient who are lactose-intolerant
* Revision surgery
* Open surgery
* Comorbidities preventing surgery
* Patients with a history of mania, depression, or schizophrenia
* Patients taking any of the following drugs or supplements

  * Anticholinergic agents
  * Benzodiazepines
  * Central nervous system depressants
  * Droperidol
  * Hydroxyzine
  * Levomepromazine or methotrimeprazine
  * Monoamine oxidase inhibitors
  * Ritonavir
  * Selective serotonin reuptake inhibitors
  * Sympathomimetics
  * St. John's Wort
* Current diagnosed alcohol or drug abuse
* Patients who cannot or will not abide by the medication restrictions listed below

Medication restrictions

* Participants must agree to abstain from using recreational or medical marijuana products or cannabidiol (CBD) in any form during the treatment period
* Participants should not drink alcohol or take other drugs while taking the study drug or hydrocodone/acetaminophen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | up to 7 days post-surgery
  Count of number of hydrocodone/acetaminophen tablet consumed

SECONDARY OUTCOMES:
Pain Visual Analog Scale (VAS) | up to 7 days post-surgery
  Scored from 0 (no pain) to 10 (worst possible pain)
Patient-Reported Outcomes Measurement Information System (PROMIS) Bank v1.1 - Pain Interference | up to 21 days post-surgery
  PROMIS measures generate T-scores. T-scores are standard scores with a mean of 50 and standard deviation of 10 in a reference population (usually U.S. general population). A low score indicates less pain interference (better outcome) and a high score indicates more pain interference (worse outcome).
PROMIS Bank v2.0 - Pain Behavior | up to 21 days post-surgery
  PROMIS measures generate T-scores. T-scores are standard scores with a mean of 50. A low score indicates less pain (better outcome) and a high score indicates more pain (worse outcome).
PROMIS Bank v2.0 - Physical Function | up to 21 days post-surgery
  PROMIS measures generate T-scores. T-scores are standard scores with a mean of 50. A low score indicates worse physical functioning and a high score indicates better physical functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Vehniah K Tjong, MD, Principal Investigator — Northwestern Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States